CLINICAL TRIAL: NCT06581237
Title: The Effects of App-Based Dietary Guidance on Determinants of Underfueling and Performance in Female Collegiate Soccer Players
Brief Title: Nutrition for Health and Performance in Female Collegiate Soccer Players
Acronym: Eat2Win-CWRU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20240738
Record Dates: First submitted 2024-08-07; First posted 2024-09-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: relative energy deficiency in sport (RED-S); performance; health; nutrition; dietetics; eHealth
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eat2Win App (Experimental): Participants will be provided a sport-specific nutrition program on the Eat2Win app.
  Interventions: Other: Eat2Win App

INTERVENTIONS:
Other: Eat2Win App — Voluntary use of the app will occur throughout the sport season.

SUMMARY:
The purpose of this research study is to conduct a pilot trial using an app-based approach to improve the health and performance of female collegiate soccer athletes through nutrition education and personalized feedback. The app-based program is designed to promote better performance through education on sport-specific fueling and good nutrition practices.

DETAILED DESCRIPTION:
Objectives: Combat female soccer athletes underfueling during their competitive season.

Study Overview: This project proposes an open label, pilot research endeavor between the Department of Nutrition at Case Western Reserve University (CWRU), Pennington Biomedical Research Center (PBRC) and the NCAA Division III CWRU Women's Soccer Team. The proposed study design will implement a commercially available, dietitian-designed phone app, Eat2Win. Eat2Win provides targeted nutritional education, specifically for soccer athletes, to improve fueling for sport and health. Additionally, Eat2Win's photo-based phone app technology will be used to provide individualized feedback to improve athlete fueling. Anthropometric, aerobic fitness (VO2), resting metabolic rate, physical activity, body composition and health-related questionnaire data will be collected from a subset of athletes at three timepoints: pre-season, in-season, and post-season. Biological measures from fingerstick blood and breath will be collected in a subset of participants at the three timepoints.

General Aims/Hypothesis: Our intervention will strive to improve athlete health and performance through nutrition education and personalized feedback using the Eat2Win app.

ELIGIBILITY:
Inclusion Criteria:

* Currently active and NCAA-eligible (including academic standing) member of the Case Western Reserve University (CWRU) Women's Soccer Team
* Owns a mobile device compatible with the Eat2Win Dietary App platform
* Signed Informed Consent

Exclusion Criteria:

* Pregnant women or women who are nursing
* Unwilling to provide anthropometric and/or biological (i.e. finger prick blood) samples during collection periods
* History of diagnosed disordered eating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Low Energy Availability in Females Questionnaire (LEAF -Q) | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Focuses on physiological symptoms of insufficient energy intake. includes 25 questions arranged in three separate, sequential sections: injuries, gastrointestinal, and reproductive functions. (score; 0-36; total score ≥8 is to be considered at risk)

SECONDARY OUTCOMES:
Resting Energy Expenditure | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Indirect calorimetry-determined resting energy expenditure expressed as kilocalories per day and adjusted for the residual difference between measured and predicted values determined as a function of fat mass, fat-free mass, age and sex according to best practices in the field.
Grip Strength | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Grip force in kilograms determined by a handgrip dynamometer, conducted on both arms, according to standard practice procedures.
Contextual Body Image Questionnaire for Athletes (CBIQA) | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Measures four dimensions of body image (Appearance (3 questions), Body Shape (3 questions), Muscularity (3 questions) and Body Weight and Fat (5 questions)) in the context of both athletics and daily life. (7-point Likert scale for each question; scaled scores for each of the four dimensions are obtained by dividing the sum of each question score within that dimension divided by the number of questions in that dimension; scoring is relative to each question with a score of 4 being neutral)
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Measures eating disorder psychopathology. It provides a measure of the range and severity of eating disorder features. (score; continuous beginning at 0; a higher score means greater risk)
Body Composition - Fat Mass | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Fat mass (kilograms) and as a percent of total body mass.
Body Composition - Fat Free Mass | Baseline/Pre-season (August 2024), Mid-season (~2 months after baseline; October 2024), End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Fat Free Mass (kilograms) and expressed as a percent of total body mass.

OTHER OUTCOMES:
Breath Analysis | Baseline/Pre-season (August 2024) and End of Study/End of Competitive Season (~4 months after baseline; December 2024)
  Untargeted gas chromatography tandem mass spectrometry analysis of breath molecules. (semi-quantitative; parts per million and parts per billion)
Eat2Win App Use - Usage Time | up to 4 months after baseline; December 2024
  Usage of the Eat2Win app during the course of the study. Presented as app usage time (hours:minutes).
Eat2Win App Use - App Clicks | up to 4 months after baseline; December 2024
  Usage of the Eat2Win app during the course of the study. Presented as clicks (number) within the app for utilizing app functions.
Eat2Win App Use - App Scoring | up to 4 months after baseline; December 2024
  Usage of the Eat2Win app during the course of the study. Presented as a numerical score within the app for utilizing app functions.
Total Energy Nutritional Intake | Collected weekly during the study, about 4 months from Baseline to End of Study Visits.
  Total Energy (kcals) quantified by the automated self-administered 24-hour dietary assessment tool.
Protein Nutritional Intake | Collected weekly during the study, about 4 months from Baseline to End of Study Visits.
  Protein Nutritional Intake (grams) quantified by the automated self-administered 24-hour dietary assessment tool.
Carbohydrate Nutritional Intake | Collected weekly during the study, about 4 months from Baseline to End of Study Visits.
  Carbohydrate Nutritional Intake (grams) quantified by the automated self-administered 24-hour dietary assessment tool.
Fat Nutritional Intake | Collected weekly during the study, about 4 months from Baseline to End of Study Visits.
  Fat Nutritional Intake (grams) quantified by the automated self-administered 24-hour dietary assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Kristyen Tomcik, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request, with appropriate data sharing agreements in place, and according to institutional policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: https://case.edu/research/compliance/human-research-protection-program/cwru-institutional-review-board